CLINICAL TRIAL: NCT06498206
Title: Dichoptic Augmented Reality (AR) Training Versus Patching for Unilateral Amblyopia in Children and Adults
Brief Title: AR Training Versus Patching in Unilateral Amblyopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other); Shanghai Tongren Hospital, Shanghai Jiao Tong University School of Medicine (Unknown); Jiangsu Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-ARTA
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Amblyopia Unilateral
Keywords: Augmented reality training; Dichoptic therapy; Patching

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AR training group (Experimental): Dichoptic augmented reality training with dual-pathway (parvocellular pathway and magnocellular pathway) and interocular push-pull paradigms developed based on neural deficits in unilateral amblyopia.
  Interventions: Other: AR training
- Patching group (Active Comparator): Conventional patching therapy.
  Interventions: Other: Patching

INTERVENTIONS:
Other: AR training — Dichoptic augmented reality training with dual-pathway (parvocellular pathway and magnocellular pathway) and interocular push-pull paradigms developed based on neural deficits in unilateral amblyopia.
  Arms: AR training group
Other: Patching — Conventional patching therapy.
  Arms: Patching group

SUMMARY:
This is a multi-center, randomized controlled trial to compare the effectiveness of AR training with patching for the treatment of unilateral amblyopia.

Specific Aim 1 (Primary): To compare the improvement of visual acuity in the amblyopic eye between AR training and patching for the treatment of unilateral amblyopia.

Specific Aim 2 (Secondary): To compare the improvement of visual functions between AR training and patching for the treatment of unilateral amblyopia.

DETAILED DESCRIPTION:
Poor compliance, limited improvement of visual functions, and regression after recovery of visual acuity have been observed in the management of amblyopia using conventional patching. Recently, dichoptic/binocular digital therapy has been developed, but no widely accepted binocular treatments with superiority available for children and adults with amblyopia (Pineles et al., 2020; Oscar et al., 2023). Here, we designed an innovative binocular therapy using augmented reality (AR) training, based on neural deficits in amblyopia, to achieve better outcomes.

Selective deficits were found in the parvocellular pathway (P pathway) compared to the magnocellular pathway (M pathway) in the monocular processing of visual information in the amblyopic eye (AE) (Wen et al., 2021). In addition to monocular deficits, imbalanced binocular suppression may also play important roles in the visual deficits of amblyopia as suggested by clinical evidence (DeSantis, 2014; Von Noorden, 1996) and psychophysical studies (Baker et al., 2008; Holopigian et al., 1988; Li et al., 2011; Zhou et al., 2013). Based on the neural deficits in unilateral amblyopia, we first apply the push-pull approach (Xu, He & Ooi, 2010; Ooi et al., 2013), which was aimed to reduce sensory eye dominance in previous literatures, into the rebalance of functions of M and P pathways in the AE and the rebalance of binocular interaction, to improve the high spatial detail perception of the AE in daily life under binocular viewing condition, as well as binocular functions.

Using AR technique combined with dichoptic device, we present differentially-processed images to each eye of the patients in real time, allowing them to interact with the surrounding environment during the visual training. Using a Butterworth filter with the cutoff at 2 cycle pre degree, the images captured in real time are divided into information with high and low spatial frequencies (SFs) corresponding to the P and M pathways, respectively. For the AE, original low SF phase of captured images is scrambled into random noise with the refresh rate of the display, while the original information with high SF is retained completely. As a result, the function of the P pathway is pulled while the function of the M pathway is pushed, actively encouraging the interaction with the surrounding environment through high SF information. For the fellow eye (FE), original high SF phase of captured images is scrambled into random noise with increased contrast and reduced temporal frequency, while the contrast of the original high SF information is reduced. As a result, in addition to the push-pull in monocular P&M pathways, the function of the P pathway in the FE is pulled and while the function of the P pathway in the AE is pushed, actively improving the rebalance of binocular inhibition.

The proposed trial will be conducted in 4 different study sites in China. For the AR training group, patients need to perform AR training for 2 hours per day at home. For the patching group, patients need to patch the FE for 2 hours per day at home.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 5-55 years (including 5 years and 55 years);
2. Best-corrected visual acuity worse than 20/30 but no worse than 20/200 in the amblyopic eye, interocular difference of 2 or more lines, with the better eye within the normal range;
3. Patients have applied optical refractive correction for more than 3 months;
4. Ability attend visits and complete the treatment;
5. Normal binocular alignment including strabismic amblyopia with orthotropia after surgical correction, or intermittent exotropia within a range of -15 to 0 prism diopters measured by the prism cover test.

Exclusion Criteria:

1. Organic eye diseases preventing the establishment of good vision (e.g. ptosis, media opacity, nystagmus, paracentral fixation, acute inflammation like keratitis, optic nerve diseases like glaucoma, retinal diseases);
2. Lesions of the brain preventing the establishment of good vision (e.g. cortical visual impairment);
3. Implantable electronic device;
4. A history of ocular surgery (except strabismus surgery) affecting vision (e.g. retinal detachment repair);
5. A history of ocular trauma affecting vision;
6. Receiving amblyopia therapy (except wearing glasses) within 2 weeks prior to presentation;
7. History of epilepsy or mental illness, or cognitive defects;
8. Currently taking medications or needing to take medications during the study period that may affect vision;
9. Inability to comply with the treatments or follow-up visits required;
10. Participation in clinical trials on drugs within 3 months prior to presentation, or clinical trials on other medical devices within 30 days prior to presentation.

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total effective rate | 13 weeks
  The effective rate is defined as the proportion of patients whose best-corrected visual acuity (BCVA) at distance improved ≥0.2 LogMAR after treatment compared to the baseline. BCVA at distance is measured with ETDRS chart.

SECONDARY OUTCOMES:
Change in best-corrected visual acuity | 2 weeks, 4 weeks, 9 weeks, 13 weeks
  Best-corrected visual acuity is measured with cycloplegic refraction, using ETDRS chart.
Effective rate | 2 weeks, 4 weeks, 9 weeks
  The effective rate is defined as the proportion of patients whose best-corrected visual acuity (BCVA) at distance improved ≥0.2 LogMAR after treatment compared to the baseline. BCVA at distance is measured with ETDRS chart.
Change in habitual visual acuity | 2 weeks, 4 weeks, 9 weeks, 13 weeks
  Habitual visual acuity is measured under habitual refractive correction at a viewing distance of 4 meters, using ETDRS chart.
Change in stereopsis | 2 weeks, 4 weeks, 9 weeks, 13 weeks
  Near and far stereopsis measured with Randot Stereotest pattern.
Change in contrast sensitivity | 2 weeks, 4 weeks, 9 weeks, 13 weeks
  Contrast sensitivity in each eye measured with contrast sensitivity testing instrument CSV-1000®.
Compliance rate | 2 weeks, 4 weeks, 9 weeks, 13 weeks
  Compliance rate is measured by daily card in the patching group and by background recording in the AR training group.
  Compliance Rate (%) = (Completed Treatment Days / Scheduled Treatment Days) × 100
Safety reports | 2 weeks, 4 weeks, 9 weeks, 13 weeks
  Assessment of the types (adverse event, serious adverse event, device deficiency), incidence rate (%), and frequency (number of events) of adverse events and device-related adverse events occurring during the clinical trial.

OTHER OUTCOMES:
Normal proportion in the worth-4 dot test | 2 weeks, 4 weeks, 9 weeks, 13 weeks
  The proportion of patients in each group with normal results in the worth-4 dot test.
Normal proportion in the Bagolini striated glasses test | 2 weeks, 4 weeks, 9 weeks, 13 weeks
  The proportion of patients in each group with normal results in the Bagolini striated glasses test.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
We concerns about patient privacy issues and it's better to protect the publication potential.

REFERENCES:
- [Background] Pineles SL, Aakalu VK, Hutchinson AK, Galvin JA, Heidary G, Binenbaum G, VanderVeen DK, Lambert SR. Binocular Treatment of Amblyopia: A Report by the American Academy of Ophthalmology. Ophthalmology. 2020 Feb;127(2):261-272. doi: 10.1016/j.ophtha.2019.08.024. Epub 2019 Oct 13. PMID 31619356
- [Background] Cruz OA, Repka MX, Hercinovic A, Cotter SA, Lambert SR, Hutchinson AK, Sprunger DT, Morse CL, Wallace DK; American Academy of Ophthalmology Preferred Practice Pattern Pediatric Ophthalmology/Strabismus Panel. Amblyopia Preferred Practice Pattern. Ophthalmology. 2023 Mar;130(3):P136-P178. doi: 10.1016/j.ophtha.2022.11.003. Epub 2022 Dec 14. No abstract available. PMID 36526450
- [Background] Wen W, Wang Y, Zhou J, He S, Sun X, Liu H, Zhao C, Zhang P. Loss and enhancement of layer-selective signals in geniculostriate and corticotectal pathways of adult human amblyopia. Cell Rep. 2021 Dec 14;37(11):110117. doi: 10.1016/j.celrep.2021.110117. PMID 34910903
- [Background] DeSantis D. Amblyopia. Pediatr Clin North Am. 2014 Jun;61(3):505-18. doi: 10.1016/j.pcl.2014.03.006. Epub 2014 Apr 14. PMID 24852148
- [Background] Von Noorden GK. Binocular vision and ocular motility. Theory and Management of Strabismus. 1996.
- [Background] Baker DH, Meese TS, Hess RF. Contrast masking in strabismic amblyopia: attenuation, noise, interocular suppression and binocular summation. Vision Res. 2008 Jul;48(15):1625-40. doi: 10.1016/j.visres.2008.04.017. Epub 2008 Jun 10. PMID 18547600
- [Background] Holopigian K, Blake R, Greenwald MJ. Clinical suppression and amblyopia. Invest Ophthalmol Vis Sci. 1988 Mar;29(3):444-51. PMID 3343099
- [Background] Li J, Thompson B, Lam CS, Deng D, Chan LY, Maehara G, Woo GC, Yu M, Hess RF. The role of suppression in amblyopia. Invest Ophthalmol Vis Sci. 2011 Jun 13;52(7):4169-76. doi: 10.1167/iovs.11-7233. PMID 21447685
- [Background] Zhou J, Huang PC, Hess RF. Interocular suppression in amblyopia for global orientation processing. J Vis. 2013 Apr 22;13(5):19. doi: 10.1167/13.5.19. PMID 23608341
- [Background] Xu JP, He ZJ, Ooi TL. Effectively reducing sensory eye dominance with a push-pull perceptual learning protocol. Curr Biol. 2010 Oct 26;20(20):1864-8. doi: 10.1016/j.cub.2010.09.043. Epub 2010 Oct 14. PMID 20951044
- [Background] Ooi TL, Su YR, Natale DM, He ZJ. A push-pull treatment for strengthening the 'lazy eye' in amblyopia. Curr Biol. 2013 Apr 22;23(8):R309-10. doi: 10.1016/j.cub.2013.03.004. PMID 23618663
- [Derived] Zhou Y, Guo S, Ling L, Gao Y, Duan X, Liu Y, Liu R, Liu H, Wang H, Lin J, Zhao C, Zhang P, Wen W. Efficacy and safety of augmented-reality pathway-specific binocular training in patients with unilateral amblyopia (ARPSBT): study protocol for a multicenter randomized controlled trial. Trials. 2025 Jul 1;26(1):232. doi: 10.1186/s13063-025-08927-2. PMID 40598549